CLINICAL TRIAL: NCT04368702
Title: Clinical Onboard Utilization of Image Guided Radiation Therapy With Magnetic Resonance (CONFIRM): A Master Protocol
Brief Title: CONFIRM: Magnetic Resonance Guided Radiation Therapy
Acronym: CONFIRM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Raymond Mak, Principal Investigator, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-665
Record Dates: First submitted 2020-04-22; First posted 2020-04-30 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Gastric Cancer; Invasive Breast Cancer; in Situ Breast Cancer; Mantle Cell Lymphoma; Larynx Cancer; Bladder Cancer
Keywords: Gastric Cancer; Invasive Breast Cancer; in Situ Breast Cancer; Lymphoma; Larynx; Bladder
MeSH Terms: conditions — Stomach Neoplasms; Breast Carcinoma In Situ; Lymphoma, Mantle-Cell; Laryngeal Neoplasms; Urinary Bladder Neoplasms; Lymphoma; Laryngeal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (5):
- Phase I - Gastric Cancer (Experimental): The research study procedures include:
  * Screening for eligibility
  * Study treatment including evaluations
  * MR-image guided radiation will be administered per disease site standards.
  * Follow up visits
  * Questionnaires
  Interventions: Radiation: Viewray MRIdian® Linac
- Phase I - Breast Cancer (Experimental): The research study procedures include:
  * Screening for eligibility
  * Study treatment including evaluations
  * MR-image guided radiation will be administered per disease site standards.
  * Follow up visits
  * Questionnaires
  Interventions: Radiation: Viewray MRIdian® Linac
- Phase I - Mantle Cell Lymphoma (Experimental): The research study procedures include:
  * Screening for eligibility
  * Study treatment including evaluations
  * MR-image guided radiation will be administered per disease site standards.
  * Follow up visits
  * Questionnaires
  Interventions: Radiation: Viewray MRIdian® Linac
- Phase I - Larynx (Experimental): The research study procedures include:
  * Screening for eligibility
  * Study treatment including evaluations
  * MR-image guided radiation will be administered per disease site standards.
  * Follow up visits
  * Questionnaires
  Interventions: Radiation: Viewray MRIdian® Linac
- Phase I - Bladder (Experimental): The research study procedures include:
  * Screening for eligibility
  * Study treatment including evaluations
  * MR-image guided radiation will be administered per disease site standards.
  * Follow up visits
  * Questionnaires
  Interventions: Radiation: Viewray MRIdian® Linac

INTERVENTIONS:
Radiation: Viewray MRIdian® Linac — MR-image guided radiation will be administered per disease site standards.

SUMMARY:
This research is being done to determine the safety and feasibility of using a type of radiation guided by magnetic resonance imaging (MRI) and chemotherapy to treat patients with gastric and breast cancer. The name of the radiation machine involved in this study is the MRIdian Linear Accelerator.

DETAILED DESCRIPTION:
This is a master clinical protocol evaluating magnetic resonance (MR) image guided radiation in patients with gastric and breast cancer.

In this research study, the investigators are researching if getting an MRI during radiation is a feasible way to delivery radiation. In this research study, a MRI done during treatment will help doctors adapt the radiation to target the most precise spot where the cancer is located.

The research study procedures include:

* Screening for eligibility
* Study treatment including evaluations
* Follow up visits
* Questionnaires

This is a Phase I/II clinical trial. A Phase I clinical trial tests the safety of investigational radiation treatment and also tries to define the appropriate dose of the investigational radiation treatment to use for further studies. "Investigational" means that the way the radiation treatment is delivered is being studied.

This research study is a Feasibility Study, which means it is the first-time investigators at this institution are examining this type of MR-guided radiation. Investigators at other hospitals and academic centers are already using this type of radiation.

The U.S. Food and Drug Administration (FDA) has approved this radiation machine and these drugs as treatment options for gastric and breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed malignancy requiring radiation
* Age 18 years of older
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* Ability to understand and the willingness to sign a written informed consent document.
* Any further criteria listed in the specific disease site cohort

Exclusion Criteria

* History of allergic reactions attributed to gadolinium-based IV contrast

  -- Note: If patient will not receive contrast, this is not applicable and kidney function will not affect eligibility
* Severe claustrophobia or anxiety
* Participants who cannot undergo an MRI
* Any other exclusion criteria listed in the specific disease site cohort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2029-06-18 (Estimated); Study Completion 2029-06-18 (Estimated)

PRIMARY OUTCOMES:
Number of Patients and delivering MR-image guided radiation-Phase I | 5 weeks
  Master feasibility study evaluating MR-image guided radiation. Feasibility is defined as Enrolling patients and delivering MR-image guided radiation on the MR Linac
Tumor Assessment with MR Guidance-Phase I | 5 weeks
  Master feasibility study evaluating MR-image guided radiation. Feasibility is defined as assessing tumor using MR guidance before, during and after MR-guided treatment patient.
Patient reported outcomes (PROMs) -Phase II | 1 year
  PROMs are collected at patient visits. PROMs will be evaluated using the Patient-Reported Outcomes Measurement Information System (PROMIS). The PROMIS Global-10 metric collects information on symptoms and quality of life.
1-year tumor control-Phase II | 1 year
  Tumor response 1 year after radiation treatment
Rate of Pathologic complete response-Gastric | 1 year
  full pathological review of surgical specimen according to the AJCC Staging Classification, 8th edition. pCR will be defined as the absence of any viable tumor cells within the pathologic specimen.

SECONDARY OUTCOMES:
Number of Participants with Treatment Related Adverse Events as Assessed CTCAE version 5.0. | 90 Days
  Toxicity of MRgRT with concurrent chemotherapy will be summarized by category and grade according to CTCAE version 5.0.
Number of Participants with Treatment Related Adverse Events as Assessed CTCAE version 5.0. | 1 year
  CTCAE version 5.0.
Duration of treatment with goal of >80% of cases treated within 90 minutes | 7 weeks
  Total time of treatment for each fraction
Number of treatment fractions that would have resulted in unacceptably high dose (exceeding constraint) to an OAR without MR-image guided radiation. | 5 Weeks
  Importance of MR-guidance
Progression Free Survival | irst date of protocol therapy to the earliest date of disease progression per RECIST criteria or death due to any cause up to 12 Months
  Estimated using the Kaplan Meier method with 95% confidence intervals based on the complementary log-log transformation.
Overall Survival | irst date of protocol therapy to the date of death due to any cause. OS time will be censored at the date of last follow-up for patients still alive up to 1 year
  The OS rate will be estimated using the Kaplan-Meier method with 95% confidence intervals based on the complementary log-log transformation.
Characterizing MRI-based tumor alterations/changes following MR-image guided radiation | 1 Year
  Evaluation of tumor response following treatment

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Mak, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu